CLINICAL TRIAL: NCT04436575
Title: Interest of Clinical Ultrasound in Patients Consulting for Acute Gastrointestinal Bleeding in the Emergency Department: an Observational Monocentric Study
Brief Title: Point-of-care Ultrasound Interest in Acute Gastrointestinal Bleeding Emergency Department Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SUD Association pour le Développement de la Recherche et de lEnseignement (Other)
Responsible Party: Principal Investigator, Thibaut MARKARIAN, Principal Investigator, SUD Association pour le Développement de la Recherche et de lEnseignement
Other Study IDs: TMarkarian/Ecuhda
Record Dates: First submitted 2020-05-21; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Acute Gastrointestinal Bleeding
Keywords: emergency department; acute gastrointestinal bleeding; echocardiography
MeSH Terms: conditions — Emergencies | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Point-of-care ultrasound — Point-of-care ultrasound prognostic performance : echocardiography mainly
  Other Names: Echocardiography

SUMMARY:
Acute Gastrointestinal (GI) Bleeding are a common chief complaint among Emergency Department. The mortality rate for Lower GI Bleeding is 3.9%. While the mortality rate can be as high as 10% for Upper GI Bleeding. Most existing scores take into account hemodynamic parameters such as systolic blood pressure or heart rate. Studies have shown that hemodynamic instability only develops late in the course of a bleed, as evidenced by a blood depletion of 30 to 40% of the total blood volume. Currently, few studies have examined the value of echocardiography in the management of patients presenting for Acute GI Bleeding in the Emergency Department. The main objective of this study is to show whether simple ultrasound parameters can, combined with clinico biological parameters, predict in an early manner the evolution of the patient presenting to the Emergency Department for Acute Gastrointestinal Bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Primary reason for emergency Department admission is acute gastrointestinal bleeding

Exclusion Criteria:

* Pregnant or breastfeeding women
* Persons not benefiting from a social security scheme
* Persons deprived of liberty
* Patient participates in another study
* The patient is in a period of exclusion determined by a previous study.
* The patient is under legal protection, guardianship or trusteeship.
* Patient refuses to participate
* It proves impossible to give informed information about the subject matter
* The patient is not fluent in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed in investigative emergency department whose primary reason for management is acute gastrointestinal bleeding may be included. Patients with echocardiography are included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of ultrasound parameters with the occurrence of adverse events | 1 day
  The primary outcome was to determine the correlation of echocardiography parameters to detect adverse events (AEs). Echocardiography parameters included signs of severe hypovolemia (end systolic left ventricular obliteration and/or complete inspiratory collapse of the inferior vena cava and/or E velocity < 0.7 m/s). Adverse events were defined as blood transfusion, therapeutic intervention to control haemorrhage (endoscopic, radiologic or surgical hemostasis), rebleeding and in-hospital mortality.

SECONDARY OUTCOMES:
Echocardiography and clinical scores | 1 day
  Correlation of echocardiographic signs of severe hypovolemia (end systolic left ventricular obliteration and/or complete inspiratory collapse of the inferior vena cava and/or E velocity < 0.7 m/s) with existing clinical scores (Glasgow-Blatchford bleeding score and Rockall score).
  The Glasgow-Blatchford bleeding score includes measurements of hemoglobin in grams per deciliter, blood urea nitrogen in millimoles per liter, initial systolic blood pressure in millimeters of mercury, sex, heart rate in beats per minute, melena present, recent syncope, hepatic disease history and cardiac failure present.
  The Rockall score includes measurement of age, shock present, comorbidities, diagnosis and major stigmata of recent hemorrhage.
Other ultrasound parameters with the occurrence of adverse events | 1 day
  The correlation of other echocardiography parameters (visual assess of the ejection fraction (in percentage) and E/A ratio (represents the ratio of peak velocity blood flow from left ventricular relaxation in early diastole = the E velocity in meter per second, to peak velocity flow in late diastole caused by atrial contraction = the A velocity in meter per second) and E' velocity (in centimeter per seconds) and ratio E/E' (ratio between early mitral inflow velocity = the E velocity in centimeter per second and mitral annular early diastolic velocity = the E' velocity in centimeter per second) and subaortic velocity time index (VTI in centimeter) with the occurrence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- MARKARIAN Thibaut, Marseille, France

IPD SHARING:
Plan to Share IPD: No